CLINICAL TRIAL: NCT06990074
Title: An Early Feasibility, Prospective, Single-Arm Study of the Polaris System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Horizon Surgical Systems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-001
Record Dates: First submitted 2025-05-06; First posted 2025-05-25 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cataract, Age-Related
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Participants with age-related uncomplicated cataract (Experimental): Single eye cataract robot-assisted cataract surgery.
  Participants will receive intraoperative eye preparation according to the standard of care for cataract surgery. Under general anesthesia, a docking procedure between the study eye and the medical device will be completed. The surgeon will use the Polaris System to perform initial surgical tasks and perform the initial portion of the affected lens extraction. Finally, the surgeon will use the Polaris System to complete the lens extraction and perform the final surgical tasks, including the intraocular lens implantation.
  Interventions: Device: cataract surgery

INTERVENTIONS:
Device: cataract surgery — Robot-assisted cataract surgery
Device: cataract surgery — Robot-assisted cataract surgery, designed to provide superior precision and increase the safety profile of the current standard of care.

SUMMARY:
A multicenter, single-arm, prospective, non-randomized, non-masked study.

DETAILED DESCRIPTION:
The study aims to assess the safety of the Polaris System in assisting surgeons to perform cataract surgery.

The Polaris System is intended to enhance precision and safety over the current standard of care by employing improved stability controls and augmented visualization properties, enabling safer surgical decisions and finer control of surgical instruments.

This study will be conducted at up to 3 research sites. After the informed consent process, potential participants will be considered enrolled in the study and undergo the screening evaluation. Following confirmation of eligibility, selected participants will be sequentially assigned to undergo robot-assisted cataract surgery and receive four scheduled follow-ups over 90 days, post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 40 and 75 (inclusive) years of age (measured at baseline)
* A slit-lamp diagnosis of uncomplicated, age-related visually significant cataract that is not posterior polar or congenital
* Eligible to undergo cataract extraction by phacoemulsification with intraocular lens (IOL) implantation
* Able and willing to comply with all study procedures
* Able to return for scheduled follow-up examinations
* Willing to adhere to the prescribed medication regimen (to prevent inflammation and infection)
* Provision of signed and dated informed consent form

Exclusion Criteria:

* Contraindication to general anesthesia
* Posterior polar or congenital cataract
* Previous history of vitrectomy, corneal, refractive, or cataract surgery
* Concurrent participation in another ophthalmological clinical study
* Allergies to any medications required in surgery, pre- and post-operative treatment
* Diagnosis of corneal disease or pathology that precludestransmission of optical coherence tomography (OCT) laser wavelength (e.g., corneal opacity), distorts OCT laser light (e.g., corneal scarring or history of radial keratotomy), or compromises engagement of the patient interface (e.g., megalocornea or pterygium), in the opinion of the Investigator
* History of poor pupil dilation, demonstration of poor reaction to pupil-dilation drugs (minimum 7 mm dilation should be targeted for study), diagnosis of a pupillary defect that precludes the iris from adequate peripheral retraction, and/or diagnosis of floppy iris syndrome or iris dyscoria
* Current or prior use of concomitant medications known to cause floppy iris syndrome (e.g., alpha-blockers, such as Flomax)
* Compromised cornea (e.g., Fuchs endothelial dystrophy)
* History of lens or zonular instability
* Immunocompromised or diagnosis of ophthalmic disease: ocular herpes zoster or simplex, lupus, collagenosis or other acute or chronic illnesses that increase the risk to the subject or confounds the outcomes of this study, in the opinion of the Investigator
* Developmental disability or cognitive impairment that would make informed consent and the assessment of visual acuity impossible, in the opinion of the Investigator
* History of significant ocular trauma
* History of iritis or uveitis
* Pregnant women, as confirmed via urine pregnancy test for women of child-bearing age at screening

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Rate of safety events | 12 weeks
  Rate of ocular adverse events in the study eye

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Quesada SA de CV, San Salvador, San Salvador Department, El Salvador

IPD SHARING:
Plan to Share IPD: No